CLINICAL TRIAL: NCT01735968
Title: A Dose-finding Phase Ib Multicenter Study of Imatinib in Combination With the Oral Phosphatidyl-inositol 3-kinase (PI3K) Inhibitor BYL719 in Patients With Gastrointestinal Stromal Tumor (GIST) Who Failed Prior Therapy With Imatinib and Sunitinib
Brief Title: A Dose-finding Study of a Combination of Imatinib and BYL719 in the Treatment of 3rd Line GIST Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571X2103; 2012-003273-25 (EudraCT Number)
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2019-09

CONDITIONS: 3rd Line GIST
Keywords: Imatinib mesylate; STI571; BYL719; GIST; 3rd line GIST
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI571 (imatinib mesylate) and BYL719 (Experimental): The study will comprise of 2 parts. A dose escalation and a dose expansion part. All patients in the dose escalation part will have a pharmacokinetic (PK) run-in period of 7 days receiving imatinib monotherapy. Patients will receive increasing doses of BYL719 (200, 300, 400 mg) in combination with 400mg imatinib daily until maximum tolerated dose (MTD) and rapid phase 2 dose (RP2D) is determined. Approximately 35 patients will enter the expansion phase.
  Interventions: Drug: ST571 + BYL719

INTERVENTIONS:
Drug: ST571 + BYL719 — Evaluable patients must meet the minimum treatment and safety evaluation requirements of the study. Patients will be treated until they experience progression of disease, withdraw consent, or experience unacceptable toxicity. One study cycle equals 28 days.

SUMMARY:
The purpose of this study is to determine a maximum tolerated dose and/or recommended phase 2 dose of a combination of imatinib and BYL719 in the treatment of 3rd line GIST patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age -WHO performance status (PS) of 0-2 -Histologically confirmed diagnosis of GIST that is unresectable or metastatic -.Available tissue specimen: • Dose-escalation part: patients must have available archival tumor tissue which can be shipped during the course of the study. In the absence of archival tumor tissue, patients must agree to a fresh pre-treatment biopsy at screening. • Dose-expansion part: patients must have available archival tumor tissue which can be shipped during the course of the study and must agree to a fresh pre-treatment biopsy
* Failed prior therapy with imatinib followed by sunitinib for the treatment of unresectable or metastatic GIST. Note the following specific criteria for the two parts of the trial: • Dose-escalation part: patients who failed prior therapy with imatinib and then have failed therapy with sunitinib. Treatment failure may be due to either disease progression on therapy (both imatinib and sunitinib) or intolerance to therapy (sunitinib) • Dose-escalation part patients may have had additional lines of therapy than imatinib and sunitinib dose-expansion part: patients must have documented disease progression on both imatinib and sunitinib. In addition, patients may have had no more than two lines of prior therapy (i.e. treatment with imatinib followed by treatment with sunitinib). • Note: Adjuvant imatinib will not count as a prior course of imatinib for the purposes of this criterion 6. Radiological (CT/MRI) confirmation of disease progression (RECIST criteria) during prior therapy with imatinib and sunitinib will be required for patients entering the Dose-expansion part

Exclusion Criteria:

-Previous treatment with PI3K inhibitors -Patient has active uncontrolled or symptomatic central nervous system (CNS) metastases Note: A patient with controlled and asymptomatic CNS metastases may participate in this trial. As such, the patient must have completed any prior treatment for CNS metastases > 28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases -Severe and/or uncontrolled concurrent medical condition that, in the opinion of the investigator, could cause unacceptable safety risks or compromise compliance with the protocol (e.g. acute or chronic liver, pancreatic disease, severe renal disease considered unrelated to study disease, chronic pulmonary disease including dyspnea at rest from any cause) -Patients with diabetes mellitus requiring insulin treatment and/or with clinical signs or with FPG >120mg/dL / 6.7mmol/L, or history of documented steroid-induced diabetes mellitus -Patient who has not recovered to grade 1 or better from any adverse events related to previous imatinib and/or sunitinib therapy before screening procedures are initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicities (DLTs) | 28 days (1st cycle)
  Dose limiting toxicity (DLT) will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) (v4.0.3), unless otherwise specified in the protocol.
Characteristics of dose limiting toxicities (DLTs) | 28 days (1st cycle)
  Dose limiting toxicity (DLT) will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) (v4.0.3), unless otherwise specified in the protocol.

SECONDARY OUTCOMES:
Frequency and characteristics of DLTs | 28 days (1st cycle)
  Dose limiting toxicity (DLT) will be assessed using CTCAE (v4.0.3), unless otherwise specified in the protocol.
Imatinib and BYL719 plasma concentrations vs time profile | 28 days (1st cycle)
Clinical benefit rate (CBR) | 28 days (1st cycle)
  Clinical benefit rate is defined as the rate of confirmed complete response (CR) or partial response (PR), or stable disease (SD) which lasts for at least 16 weeks.Tumor response will be determined locally by the investigator sites according to Novartis guideline on the Response Evaluation Criteria in Solid Tumors, based on RECIST Version 1.1.
Type of adverse drug reactions | 28 days (1st cycle)
Frequency of adverse drug reactions | 28 days (1st cycle)
Severity of adverse drug reactions | 28 days (1st cycle)
Effect of basic Pharmacokinetics (PK) parameter: AUC0-24 | 28 days (1st cycle)
Effect of basic PK parameter: Cmax | 28 days (1st cycle)
Effect of basic PK parameter: Tmax | 28 days (1st cycle)
Effect of basic PK parameter: CL/F | 28 days (1st cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Oregon Health and Science University Dept. of OHSU (3), Portland, Oregon, United States
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Bordeaux, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Candiolo, TO
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pantaleo MA, Heinrich MC, Italiano A, Valverde C, Schoffski P, Grignani G, Reyners AKL, Bauer S, Reichardt P, Stark D, Berhanu G, Brandt U, Stefanelli T, Gelderblom H. A multicenter, dose-finding, phase 1b study of imatinib in combination with alpelisib as third-line treatment in patients with advanced gastrointestinal stromal tumor. BMC Cancer. 2022 May 6;22(1):511. doi: 10.1186/s12885-022-09610-4. PMID 35524239
- See also: Results for CSTI571X2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17545